CLINICAL TRIAL: NCT02772367
Title: Generation of Induced Pluripotent Stem Cell Derived Cardiomyocytes From Patients Exposed to Trastuzumab Therapy for Breast Cancer
Brief Title: Generation of Heart Muscle Cells From Blood or Skin Cells of Breast Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: 16-025
Record Dates: First submitted 2016-05-11; First posted 2016-05-13 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: cardiotoxicity; 16-025
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — skin tissue

GROUPS / COHORTS (1):
- Breast Cancer Patients: In study participants undergoing breast reconstruction surgery prior to breast radiation therapy, we will obtain skin tissue at the time of reconstruction surgery from the surgical specimen.
  Interventions: Procedure: skin punch biopsy

INTERVENTIONS:
Procedure: skin punch biopsy

SUMMARY:
The purpose of this study is to investigate whether cells from a biopsy taken from the patient skin can be transformed into cardiomyocytes the changes in cardiomyocyte (heart muscle cells) when grown in a special culture medium outside of the body. The structure and function of these cells will then be studied to determine why some patients with breast cancer who are treated with chemotherapy including anthracycline (e.g. Doxorubicin) and anti-HER2 therapy (e.g. Herceptin) develop decreased heart function.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age greater than 18 years
* Willing to participate in protocol procedures with signed informed consent
* Assessment of LVEE via echocardiogram, cardiac MRI, or MUGA

Subjects in the cardiotoxicity group (TOX) must meet the following criteria:

* History of HER2 positive breast cancer (stage I-IV)
* Prior/current treatment with anthracycline based chemotherapy followed by anti-HER2 directed therapy or anti-HER2 directed therapy alone
* Assessment of LVEF at baseline prior to initiation of anthracycline or anti-HER2 therapy and during anti-HER2 therapy via echocardiogram, cardiac MRI, or MUGA
* Prior confirmed diagnosis of cardiotoxicity associated with anti-HER2 based therapy, defined as a decrease in LVEF > 10% from baseline to < 53% with symptoms of heart failure (NYHA class II-IV).

Subjects in the no cardiotoxicity group (NO-TOX) must meet the following criteria:

* History of HER2 positive breast cancer (stage I-IV)
* Completion of planned anthracycline and anti-HER2 therapy, or anti-HER2 therapy alone
* No symptoms of heart failure (NYHA class II-IV) during and at the end of anthracycline and anti-HER2 therapy
* Assessment of LVEF at baseline prior to innitiation of anthracycline or anti-HER2 therapy and during anti-HER2 therapy via echocardiogram, cardiac MRI, or MUGA
* Normal LVEF >53% at each assessment during and at the end of trastuzumab therapy.
* Maximum absolute decrease in LVEF <5% from baseline during and at the end of trastuzumab therapy.
* LVEF assessment performed at baseline and at least two time points during trastuzumab therapy.

Exclusion Criteria:

* Unwilling or unable to give skin biopsies
* Contraindications to punch biopsy including but not limited to bleeding diathesis, as determined by the investigator.
* Known pre-existing CV disease prior to initiation of breast cancer therapy as determined by the investigator, including

  * Obstructive coronary artery disease (stenosis >70%)
  * Arrhythmia - paroxysmal or persistent atrial arrhythmias, sustained ventricular tachycardia (>30 seconds), ventricular fibrillation, or cardiac arrest
  * Cardiomyopathy (EF <53%)
  * Heart failure (NYHA class II-IV)
  * Valvular heart disease with equal to or greater than moderate stenosis or regurgitation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan Kettering Cancer Center (MSKCC).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-05-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
derive iPSs from skin fibroblasts | 1 day
  described by Yamanaka et al with modification using the Millipore STEMCCA excisable polycystronic lentivirus reprogramming kit.2

CONTACTS AND LOCATIONS:
Overall Officials: Angel Chan, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/